CLINICAL TRIAL: NCT06366633
Title: Feasibility Open Pilot of Web-based Mind-body Treatment to Enhance Resilience Among Patients With Nontraumatic Painful Upper Extremity Conditions and Comorbid Risky Substance Use
Brief Title: Web-based Mind-body Program for Comorbid Nontraumatic Upper-extremity Condition and Risky Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jafar Bakhshaie (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Jafar Bakhshaie, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000713; 1K23AT012364-01 (NIH)
Record Dates: First submitted 2024-03-28; First posted 2024-04-16 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Orthopedic Disorder; Nontraumatic Injury; Substance Use; Upper Extremity Problem
Keywords: Upper Extremity Condition; Risky substance Use; Mindfulness; Nontraumatic conditions; Chronic pain
MeSH Terms: conditions — Musculoskeletal Diseases; Substance-Related Disorders; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-TIRELESS (Experimental): An asynchronous web-based mind-body intervention focused on decreasing disability, pain, risky substance use, and related distress in patients with nontraumatic upper-extremity conditions and comorbid risky substance use.
  Interventions: Behavioral: Web-TIRELESS

INTERVENTIONS:
Behavioral: Web-TIRELESS — This is a self-administered web-based intervention that consists of 4 30-45-minute video sessions that teach mind-body skills, cognitive-behavioral strategies (e.g., reframing, pain and substance use urge surfing), activity pacing, acceptance and commitment skills, and psychoeducation on the association between substance use and pain. The program aims to increase patients' physical and emotional functioning and decrease pain intensity and maladaptive substance use behaviors.

SUMMARY:
The investigator aims to conduct an open pilot study (N=6; 5 completers) to test the feasibility, acceptability, and credibility of an asynchronous web-based mind-body intervention (Toolkit for Resilient Life beyond Pain and Substance Use; Web-TIRELESS) for adult patients with a comorbidity of non-traumatic painful upper-extremity condition(s) (NPUC) and risky substance use.

Deliverables: 1) Adapt and refine open pilot protocol, patient recruitment, and other study materials. 2) Assess the feasibility, acceptability, and credibility of Web- TIRELESS in preparation for a future feasibility RCT.

Participants will complete 4 on-demand video sessions at their own pace (approximate pace of 1 session per week) and complete baseline and post-test assessments. participants may also partake in an exit interview to provide feedback on Web-TIRELESS to further refine the program and study protocol for future iterations.

DETAILED DESCRIPTION:
Aim: Conduct a pilot study (N=6; 5 completers) of Web-TIRELESS followed by virtual exit interviews with adult patients with painful nontraumatic upper extremity conditions and comorbid risky substance use. The investigators will use this mixed methods information to assess the feasibility, credibility, and acceptability of Web-TIRELESS and optimize the program and study methodology in preparation for a pilot feasibility randomized control trial (RCT).

The Web-TIRELESS program, adapted from the Toolkit for Optimal Recovery (P# 2020P000095), consists of 4 on-demand video sessions each being approximately 30-45 minutes long. The sessions aim to teach mind-body skills, cognitive-behavioral strategies (e.g., reframing, pain and substance use urge surfing), activity pacing, acceptance and commitment skills, and psychoeducation on the association between substance use and pain. Each session will consist of a combination of short (5-10 min) educational videos, exercises, and guided home practice goal-setting. At the end of each session, each participant will complete an interactive quiz that covers the subject of the session to facilitate deeper understanding and internalization of the session content. The interactive quiz format has been demonstrated to be useful for learning new information, including among orthopedic patients. Between sessions, participants will be encouraged to practice program skills at home. Home practice materials include Web-based audio and video clips (e.g., 5 min mindfulness of pain and substance urge). Outside the on-demand sessions, participants will continue to use the web-based platform to guide and log their home practice.

After completion of the program, participants will attend a one-time 15-30 minute exit interview to share their perceptions of Web-TIRELESS and any recommendations to improve quality. This information will be used to further adapt and optimize Web-TIRELESS prior to future study phases.

Assessments: Participants will complete baseline and post-test assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient adults seeking care in the Hand and Arm Center
2. Diagnosed with a non-traumatic painful upper-extremity condition (NPUC)
3. Pain score > 4 on the Numerical Rating Scale (NRS)
4. Risky substance use (scores >10 and <27 for alcohol, and >3 and <27 for cannabis, cocaine, amphetamine-type stimulants, inhalants, sedatives, hallucinogens, opioids, tobacco products, and e-cigarette on The World Health Organization's - Alcohol, Smoking and Substance Involvement Screening Test [WHO-ASSIST])
5. Owns a smartphone, laptop, or computer with internet access
6. Age ≥18yr
7. English fluency
8. Ability and willingness to participate in a live video focus group and the following asynchronous Web-based intervention

Exclusion Criteria:

1. Participation in mind-body or specialized substance abuse treatment in the past 3 months
2. Practice of mindfulness >45 minutes/week in the past 3 months
3. Psychotropic medications (e.g. antidepressants) changed in the past 3 months
4. Serious untreated mental illness (e.g., Schizophrenia)
5. Suicidal ideation with intent or plan
6. Pregnancy
7. Secondary gains that may bias motivation (e.g., pending disability claim),
8. Moderate to severe cognitive impairment (score ≥4 on the Short Portable Mental Status Questionnaire (SPMSQ))
9. History of surgery for the presented NPUC within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Credibility and Expectancy Questionnaire (CEQ) | Baseline (0 Weeks)
  Assesses the degree to which one believes the intervention will effectively manage their condition, substance use, and related worry. Possible scores range from 3 to 27 for both the credibility and the expectancy subscales. Higher scores represent higher credibility and expectancy.
Client Satisfaction Questionnaire to assess satisfaction with/acceptability of treatment | Post-Test (4 Weeks)
  Participant's satisfaction with treatment received after completion . The score range is 0-12. Higher scores indicate greater satisfaction.
The User Experience Scale to assess participants' satisfaction with (acceptability of) web-based delivery | Post-Test (4 Weeks)
  This measure will assess how well patients like the Wed-based program content and delivery. Total raw scores range from 22 to 110 with higher scores indicating greater satisfaction with the platform.
The percent of patients that agree to participate to assess feasibility of recruitment | Baseline (0 Weeks)
  The percent of eligible patients approached that agree to participate.
Rate at which program was accepted, measured by attendance to assess acceptability of treatment | Post-Test (4 Weeks)
  The proportion of participants who complete > or = 3 of 4 sessions.
Adherence to homework | Through intervention completion, an average of 1 month
  Rate of participant's completion of homework assigned throughout the study.
Rate of participant's completion of self-report measures to assess feasibility of assessments | Baseline (0 Weeks), Post-Test (4 Weeks)
  Investigators will report number of patients who complete assessments at each time-point.
Adverse Events | Through study completion, an average of 1 month
  Any self-reported or observed negative events related to participation

SECONDARY OUTCOMES:
Graded Chronic Pain Scale (GCPS) | Baseline (0 Weeks), Post-Test (4 Weeks)
  Assesses pain severity and pain related disability. Total scores range from 0 to 10 with high scores indicating worse pain severity.
Disabilities of the Arm, Shoulder and Hand (DASH) | Baseline (0 Weeks), Post-Test (4 Weeks)
  A 30-item measure that assesses disability severity. Scores range from 0 to 100 with higher scores indicating greater disability.
Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Depression-Short Form 8b v1.0 | Baseline (0 Weeks), Post-Test (4 Weeks)
  An 8-item measure assessing symptoms of depression. Scores range from 8 to 40 with higher scores indicating greater symptom severity
PROMIS Emotional Distress - Anxiety-Short Form 8b v1.0 | Baseline (0 Weeks), Post-Test (4 Weeks)
  An 8-item measure assessing symptoms of anxiety. Scores range from 8 to 40 with higher scores indicating greater symptom severity
Pain Catastrophizing Scale (PCS) | Baseline (0 Weeks), Post-Test (4 Weeks)
  Assesses magnification, helplessness, and rumination about pain. Scores range from 0 to 52. Higher scores indicate greater pain catastrophizing.
Pain Anxiety Symptoms Scale - Short Form (PASS-20) | Baseline (0 Weeks), Post-Test (4 Weeks)
  Assesses fear and anxiety related to pain. Scores range from 0 to 100. Higher scores indicate greater pain-related fear and anxiety.
Pain Vigilance and Awareness Questionnaire (PVAQ) | Baseline (0 Weeks), Post-Test (4 Weeks)
  Assesses preoccupation with or attention to pain. Scores range from 16 to 96. Higher scores indicate greater pain vigilance.
Brief Experiential Avoidance Questionnaire (BEAQ) | Baseline (0 Weeks), Post-Test (4 Weeks)
  This measure assesses tendencies to avoid unpleasant internal experiences. Scores range from 15 to 90. Higher scores suggest greater avoidance behaviors.
Current Opioid Misuse Measure (COMM) | Baseline (0 Weeks), Post-Test (4 Weeks)
  Assesses risk for aberrant medication-related behavior in persons with chronic pain. Scores range from 0 to 68. Higher scores indicate greater risk for opioid misuse.
The Timeline Follow Back (TLFB) | Through intervention completion, an average of 1 month
  Assesses daily estimates of alcohol, cannabis, cigarette, and other drug use during the past week. The range is 0 to 7 days, with higher scores indicating more severe use.
Numerical Rating Scale (NRS) | Baseline (0 Weeks), Post-Test (4 Weeks)
  Severity of participant's pain at rest and with activity using a Likert scale with 0 being no pain and 10 being worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jafar Bakhshaie, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital (MGH), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levey N, Chen N, Ditre J, Sylvia L, Mudgal C, Bhashyam A, Garg R, Ring D, Vranceanu AM, Bakhshaie J. A Web-Based Mind-Body Intervention to Improve Resilience Among Patients With Nontraumatic Painful Upper-Extremity Conditions and Comorbid Risky Substance Use: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2024 Dec 9;13:e64547. doi: 10.2196/64547. PMID 39652859